CLINICAL TRIAL: NCT02562612
Title: Ascending Multi-Dose Clinical Trial to Assess the Pharmacokinetics Efficacy of SM-88 Oral Administration in Breast Cancer Subjects
Brief Title: Study of SM-88 in Advanced Cancers
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was never initiated. Never established sites or enrolled subjects.
Sponsor: Tyme, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM-88-001
Record Dates: First submitted 2015-09-26; First posted 2015-09-29 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — racemetyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SM-88 (Experimental): SM-88 multiple ascending doses
  Interventions: Drug: SM-88

INTERVENTIONS:
Drug: SM-88 — Daily SM-88 in multiple ascending doses over 6 months

SUMMARY:
The purpose of this study is to collect response and pharmacokinetic data on the oral administration of a cocktail combination of 4 drugs being developed for the indication of metastatic breast cancer.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to assess the response rate and PFS in previously treated breast cancer patients. Additional objectives include the pharmacokinetics of multiple ascending doses of SM-88, a cocktail combination of 4 drugs being developed for the indication of metastatic breast cancer. Secondary objectives of this study include an assessment of safety and tolerability of ascending doses of orally administered SM-88. Additional response data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects, between 18 and 70 years of age, that are willing and able to give written informed consent.
2. Subjects must be willing and able to comply with the clinical trial procedures and timelines as outlined in the Time and Events Table.
3. Subjects should be continuous nonsmokers and have not used nicotine-containing products for at least three months prior to dosing on Day 1.
4. Body mass index (BMI) between 20 and 29.
5. As outlined in section 5.1.1.1, subjects of childbearing potential must agree to use an approved method of contraception for the duration of the clinical trial and for three months after the dose of the IMP.
6. Must be able to swallow and retain oral medication.
7. Subjects must be willing to discontinue the use of any vitamins or herbal supplements seven days prior to the IMP dosing and not resume the use of these supplements until after PK sample is collected at 168h/Day 8.

Exclusion Criteria:

1. Prior medical history of any illness or injury that, in the opinion of the principal investigator (PI), that may confound the results of the clinical trial or pose an additional risk to the subject by his participation in the clinical trial.
2. Current or historic drug or alcohol abuse.
3. Unwillingness to discontinue alcohol intake for 24 hours prior to IMP dosing until the collection of the PK sample at 168-h/Day 8.
4. Subjects should not have a history of lactose intolerance.
5. Concurrent use or known history of hypersensitivity to any of the components of SM 88.
6. Clinically significant abnormal laboratory test results at screening and/or baseline visit as determined by PI.
7. Participation in another clinical trial within 30 days prior to screening.
8. Surgery within 90 days prior to dosing determined by the PI to be clinically relevant.
9. Subjects must be considered medically healthy with no clinically significant medical history.
10. Subjects cannot be taking any concomitant medications. Subjects must be willing to discontinue the use of any vitamins or herbal supplements seven days prior to the dose date of the clinical trial and remain off these supplements until the last PK sample is obtained (168h/Day 8).
11. Positive urine drug screening.
12. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6-12 months
  Response data will be collected on SM88 in breast cancer. SM88 has previously been reported to have clinical benefit in a variety of cancers (J Clin Oncol 31, 2013. suppl; abstr e22095)
PFS | 6-12 months
  PFS data will be collected on SM88 in breast cancer. SM88 has previously been reported to have clinical benefit in a variety of cancers (J Clin Oncol 31, 2013. suppl; abstr e22095)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days
  The safety of orally administered SM-88 will be assessed by collected adverse events data as determined by physical exam, laboratory parameters and subject questionnaire.
Blood concentration of SM-88 | 168 hours
  Blood sampling will be performed to establish the pharmacokinetic profile of SM-88. Time sampling will be at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5, 6, 8, 12, 48, and 168 hours post dose.